CLINICAL TRIAL: NCT07066800
Title: Verification of the Effects of a Mindfulness-based Online Training Program for Recovering From Cognitive Decline Related to Maltreatment Experiences
Brief Title: Mindfulness Intervention for Maltreatment-Related Cognitive Decline
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Chilgok Hospital (Other)
Responsible Party: Principal Investigator, Sang Won Lee, M.D., Ph.D., Kyungpook National University Chilgok Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-05-020-001
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Health Adult Subjects; Maltreament
Keywords: Mindfulness-Based Intervention; Cognitive Function; Childhood Maltreatment

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm - Mindfulness Intervention Group (Experimental): * Participants receive a 4-week online mindfulness-based training via a structured website (videos, weekly tasks).
  * Includes breathing, body scan, and walking meditation sessions
  Interventions: Behavioral: Mindfulness-Based Online Training Program
- Control Arm - Waiting List Group (No Intervention): * Participants do not receive the intervention during the initial 4 weeks.
  * Serve as a comparison group for pre-post outcomes.
  * May receive the intervention after the study period (if planned as ethical compensation).

INTERVENTIONS:
Behavioral: Mindfulness-Based Online Training Program — A 4-week web-based mindfulness program developed by the research team, designed to improve attention, emotional regulation, and mental health in adults with a history of maltreatment.
  * The intervention includes:
    * Weekly educational videos (5-10 minutes each)
    * Weekly mindfulness practice videos (5-10 minutes each)
    * Assigned home practices each week
    * Optional support via KakaoTalk channel for Q&A and participant engagement
  * Weekly themes include:
    * Breathing and muscle relaxation
    * Mindfulness breathing meditation
    * Body scan meditation
    * Mindful walking
  Arms: Experimental Arm - Mindfulness Intervention Group

SUMMARY:
The goal of this clinical trial is to examine whether an online mindfulness-based training program can help improve cognitive function including attention, emotional regulation, and mental health (such as depression and anxiety) in young adults (ages 19 to 40) who have experienced maltreatment. The main questions it aims to answer are:

* Can a 4-week online mindfulness program improve cognitive function including attention in adults with a history of maltreatment?
* Does the program reduce symptoms of depression and anxiety compared to a control group?

Researchers will compare a mindfulness training group with a waiting-list control group to see if the intervention leads to improvements in psychological and cognitive functioning.

Participants will:

* Complete psychological and cognitive assessments before and after the 4-week period
* Watch weekly online educational and mindfulness practice videos (e.g., breathing, body scan, walking meditation)
* Perform weekly mindfulness-based assignments through a study website
* Engage in optional interaction via a chat channel

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 to 40 years
* Individuals with a history of childhood maltreatment, defined as meeting at least one of the following on the Early Trauma Inventory-Short Form (ETISR-SF)

  * At least one subscale (general trauma, physical abuse, emotional abuse, sexual abuse) exceeding established cut-off scores (Plaza et al., 2011)
  * A Global score ≥ 4 on ETISR-SF
* No current or past history of major internal medical or psychiatric disorders
* Willing and able to provide written informed consent
* Able to access and use an online platform (computer or mobile device)

Exclusion Criteria:

* Intellectual disability, defined as IQ ≤ 70
* History of traumatic brain injury
* Ongoing or past (≥6 months) psychiatric treatment for a diagnosed mental disorder
* Presence of severe psychiatric symptoms impairing reality testing or basic daily functioning (Note: Individuals with mild to moderate depressive symptoms based on screening are not excluded)

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Cognitive function_self-report | Baseline and after 4 weeks
  Conner's Adult ADHD Rating Scale Korean Version (CAARS-K)
Cognitive function_Computerized | Baseline and after 4 weeks
  Comprehensive Attention Test

SECONDARY OUTCOMES:
Depressive Symptoms | Baseline and after 4 weeks
  Center for Epidemiologic Studies Depression Scale
Anxiety Symptoms | Baseline and after 4 weeks
  Generalized Anxiety Disorder-7
Emotional Regulation Difficulties | Baseline and after 4 weeks
  Difficulties in Emotion Regulation Scale
Cognitive Emotion Regulation Strategy | Baseline and after 4 weeks
  Cognitive Emotion Regulation Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook National University Chilgok Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcomes may be shared following study completion and publication of results, but only upon formal request and at the discretion of the principal investigator. Access will be granted solely for non-commercial academic research purposes and will require a data use agreement and institutional approval.